CLINICAL TRIAL: NCT04419116
Title: Faculty of Medicine, Thammasat University
Brief Title: Clinical Outcomes Between Tibial Preservation Bone Cut and Conventional Tibial Bone Cut Following Medial UKA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Thammasat University (Other)
Responsible Party: Principal Investigator, Boonchana Pongcharoen, Associated professor, Thammasat University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MTU-EC-OT-1-137/62
Record Dates: First submitted 2020-06-01; First posted 2020-06-05 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Knee Osteoarthritis; Knee Arthropathy
Keywords: mobile bearing UKA; Oxford UKA; medial knee pain
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tibial preservation bone cut (Experimental): tibial preservation bone cut following mobile bearing UKA
  Interventions: Procedure: tibial preservation bone cut
- tibial conventional bone cut (Experimental): tibial conventional bone cut following mobilebearing UKA
  Interventions: Procedure: tibial preservation bone cut

INTERVENTIONS:
Procedure: tibial preservation bone cut — tibial preservation bone cut: removing of proximal tibial less than conventional tibial bone cut with 2mm.

SUMMARY:
The mobile bearing unicompartmental knee arthroplasty has shown excellent clinical outcome and survivorship. However, some studies have shown that the patients still had medial knee pain and shown worst the clinical outcome, even though the survivorship was excellent. The medial knee pain after operation was the one cause of revision. The incidence of medial knee pain was 0%-9%. The cause of medial knee pain was overloading on the medial plateau, local inflammation, over hanging of the tibial component and overstretching of the MCL due to the application of excessive polyethylene. Therefore, the tibia in this study was cut with under resection technique for reducing the overloading on the medial tibial plateau. The purpose of this study is to compare medial knee pain between tibial bone cut preservation technique and conventional tibial bone cut technique following mobile bearing UKA.

DETAILED DESCRIPTION:
A randomized control trial study was conducted at Thammasat University hospital, Thailand. The inclusion criteria were patients with medial osteoarthritis (OA) of the knee with an Alhback score of 2, 3 and 4, who were older than 50 years of age, with a range of movement (ROM) > 90°, a varus deformity < 25°, and flexion contracture < 20° who underwent a medial mobile bearing UKA (Oxford UKA; Zimmer Biomet, Inc, Warsaw, IN, USA), performed by a single surgeon. The exclusion criteria were patients with a diagnosis of spontaneous osteonecrosis of the knee (SPONK), intraoperative anterior cruciate ligament (ACL) insufficiency, inflammatory joint disease, gout, post-traumatic arthritis, and primary PF arthritis. The patients were randomized with computer technique into 2 groups, group (gp) I, conventional tibial bone cut technique and gp II, tibial bone cut preservation technique. The baseline patient characteristics included age, sex, site, the Knee Society Score© (KSS) (knee score, pain score, and functional score), Oxford knee score (OKS), KOOS, Kujara score, body mass index (BMI), degree of varus deformity, flexion contracture, genu recurvatum, and range of motion (ROM) were recorded. The patients were followed up at 2 weeks, 6 weeks, 3months, 6months, 1 years, and annually. The VAS ofr medial knee and incidence of medial knee pain were assessed in a blinded fashion by a research assistant at each visit using VAS scale (0-10). The KSS, OKS, KOOS, and Kujara score also were recorded. At each follow-up, the patients underwent AP standing, lateral standing, skyline view, and long-leg radiographs and the component alignment, tibiofemoral angle and joint line of femur and tibia recorded.

ELIGIBILITY:
Inclusion Criteria:

* medial osteoarthritis of knee

Exclusion Criteria:

* posttraumatic arthritis
* gout
* Rheumatoid arthritis
* anterior cruciate ligament insufficiency
* osteonecrosis of knee

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
visual analog scale (VAS) for pain | 2 years
  pain at medial tibial plateau

SECONDARY OUTCOMES:
knee society score | 2 years
  The standard knee score for determining function after knee arthroplasty
Oxford knee score | 2 years
  The standard knee score for determining function after knee arthroplasty
joint forgotten score | 2 years
  The standard knee score for determining function after knee arthroplasty
knee injury osteoarthritis outcome score | 2 years
  The standard knee score for determining function after knee arthroplasty
Kujala score | 2 years
  The standard knee score for determining function after knee arthroplasty

CONTACTS AND LOCATIONS:
Overall Officials: Boonchana Pongcharoen, Study Director — faculty of medicine, Thammasat university
Locations (1):
- Boonchana Pongcharoen, Pathum Thani, Thailand

IPD SHARING:
Plan to Share IPD: No